CLINICAL TRIAL: NCT05110430
Title: In Silico Clinical Trial Comparing the Reading Accuracy of Doctors and a Deep Learning Algorithm for Detection of Metastatic Bone Disease on Bone Scintigraphy Scans.
Brief Title: Automated Detection of Metastatic Bone Disease on Bone Scintigraphy Scans
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Collaborators: Aalborg University Hospital (Other); Centre Hospitalier Universitaire de Liege (Other); University Hospital, Aachen (Other); University of Namur (Other)
Responsible Party: Sponsor
Other Study IDs: MBDDL
Record Dates: First submitted 2021-04-19; First posted 2021-11-08 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Bone Tumor
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BS-UKA: Patients who underwent bone scintigraphy scanning between 2010 and 2018 at RTWH Aachen university hospital, and had a bone scan report that indicates the presence or absence of metastatic bone disease.
  Interventions: Other: Deep learning based detection of metastatic bone disease on bone scintigraphy scans.
- BS-Namur: Patients who underwent bone scintigraphy scanning between 2010 and 2018 at Namur university hospital, and had a bone scan report that indicates the presence or absence of metastatic bone disease.
  Interventions: Other: Deep learning based detection of metastatic bone disease on bone scintigraphy scans.
- BS-Aalborg: Patients who underwent bone scintigraphy scanning between 2010 and 2018 at Aalborg university hospital, and had a bone scan report that indicates the presence or absence of metastatic bone disease.
  Interventions: Other: Deep learning based detection of metastatic bone disease on bone scintigraphy scans.

INTERVENTIONS:
Other: Deep learning based detection of metastatic bone disease on bone scintigraphy scans. — The aim is to investigate whether deep learning algorithms can detect bone metastasis with high accuracy and specificity.

SUMMARY:
Bone scintigraphy scans are two dimensional medical images that are used heavily in nuclear medicine. The scans detect changes in bone metabolism with high sensitivity, yet it lacks the specificity to underlying causes. Therefore, further imaging would be required to confirm the underlying cause. The aim of this study is to investigate whether deep learning can improve clinical decision based on bone scintigraphy scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a bone scintigraphy scan that is available with the radiologic report between 2010-2018

Exclusion Criteria:

* The lack of a bone scan, or corresponding radiologic report

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who had an indication for undergoing bone scintigraphy in any of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 2365 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The classification performance of DL algorithm compared to the ground truth | June 2021
  Reporting the performance measures (Area under the curve, accuracy, specificity..etc)

SECONDARY OUTCOMES:
Comparing the classification performance of the DL algorithm to that of physicians | June 2021
  Correctness of the diagnosis of Dr versus AI (dichotomous variable: correct versus not correct) on a subset of the validation data, using a McNemar statistical test

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Result] Ibrahim A, Vaidyanathan A, Primakov S, Belmans F, Bottari F, Refaee T, Lovinfosse P, Jadoul A, Derwael C, Hertel F, Woodruff HC, Zacho HD, Walsh S, Vos W, Occhipinti M, Hanin FX, Lambin P, Mottaghy FM, Hustinx R. Deep learning based identification of bone scintigraphies containing metastatic bone disease foci. Cancer Imaging. 2023 Jan 25;23(1):12. doi: 10.1186/s40644-023-00524-3. PMID 36698217